CLINICAL TRIAL: NCT01272401
Title: Determinants and Correlates of Physical Activity in Breast Cancer Survivors
Brief Title: Quality of Life in Breast Cancer Patients and Survivors
Status: Completed | Type: Observational
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Edward McAuley, Professor, University of Illinois at Urbana-Champaign
Other Study IDs: UIUC_IRB_10085; 1F31AG034025-01A1 (NIH)
Record Dates: First submitted 2010-07-02; First posted 2011-01-07 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients and survivors

SUMMARY:
The purpose of this study is to determine how physical activity, other lifestyle factors, and psychosocial factors are related to quality of life and other health outcomes across the breast cancer survival spectrum from diagnosis to long term survival in a nationally representative sample of breast cancer patients and survivors across a 6 month period of time.

DETAILED DESCRIPTION:
Participants in this study will be asked to sign an informed consent, wear an activity monitor (similar to a pedometer) for 7 consecutive days and complete a packet of questionnaires. The questionnaires will take about 45 minutes to complete. All materials will be sent to participants via the US Postal Service and will need to be mailed back in the provided self-addressed stamped envelopes within 2 weeks. Participants will be asked to repeat these same assessments again in 6 months. NO lab visits will be required for participation. Women from all across the U.S. who have been diagnosed with breast cancer at any point in their lives are being sought. There is no limit on time since diagnosis or treatment status.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Have received a breast cancer diagnosis and consider self a breast cancer patient or survivor
* Aged 18 years and older
* English speaking
* No limit on time since diagnosis

Exclusion Criteria:

* Under the age of 18
* Male
* Have never been diagnosed with breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community dwelling breast cancer patients and survivors
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Quality of life. Health-related quality of life will be assessed utilizing a breast cancer specific quality of life measure and global quality of life will be assessed using the satisfaction with life scale. | Baseline
Quality of life. Health-related quality of life will be assessed utilizing a breast cancer specific quality of life measure and global quality of life will be assessed using the satisfaction with life scale. | 6 months

SECONDARY OUTCOMES:
Self-efficacy for engaging in physical activity and overcoming barriers to physical activity. | Baseline
Physical activity as measured by questionnaire and 7 day accelerometry. | Baseline
Self-efficacy for engaging in physical activity and overcoming barriers to physical activity. | 6 months
Physical activity as measured by questionnaire and 7 day accelerometry. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward McAuley, PhD, Principal Investigator — University of Illinois at Urbana-Champaign

IPD SHARING:
Plan to Share IPD: No